CLINICAL TRIAL: NCT05808166
Title: A Phase II, Randomized, Observer-blinded, Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of Hecolin® in Healthy Pregnant Women Between Gestational Age 14-34 Weeks and Non-Pregnant Women of 16-45 Years Old.
Brief Title: Safety and Immunogenicity of Hecolin® in Healthy Pregnant Women
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Open Philanthropy (Other); Bill and Melinda Gates Foundation (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IVI_Hecolin_P001
Record Dates: First submitted 2023-03-07; First posted 2023-04-11 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis E Infection
Keywords: Hepatitis E infection; Hepatitis E virus; Hepatitis E vaccine; Hepatitis E in pregnancy
MeSH Terms: interventions — hecolin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pregnant participant receiving Hecolin® (Experimental): 1 (N=1,104): Pregnant participants receiving Hecolin® (n=150 immunogenicity subset).
  For Arm 1, pregnant participants will receive 2 doses of Hecolin® at a 4 weeks interval and the third dose will be administered postpartum, approximately 20 weeks after the second dose.
  Interventions: Biological: Hecolin® (Recombinant Hepatitis E Vaccine (Escherichia coli)).
- Pregnant participants receiving placebo (Placebo Comparator): Arm 2 (N=1,104): Pregnant participants receiving placebo (n= 150 immunogenicity subset).
  For Arm 2, pregnant participants will receive 2 doses of placebo at a 4 weeks interval and the third dose will be administered postpartum, approximately 20 weeks after the second dose.
  Interventions: Other: Isotonic Sodium Chloride injection
- Non-Pregnant participants receiving Hecolin® (Active Comparator): Arm 3 (N=150): Non-Pregnant participants receiving Hecolin® (n= 150 immunogenicity subset).
  For Arm 3, non-pregnant participants will receive Hecolin® at 0-1-6 months schedule.
  Interventions: Biological: Hecolin® (Recombinant Hepatitis E Vaccine (Escherichia coli)).

INTERVENTIONS:
Biological: Hecolin® (Recombinant Hepatitis E Vaccine (Escherichia coli)). — Hecolin® will be administered 2 doses administered 4 weeks apart during pregnancy and 1 dose administered after delivery at least 20 weeks following the second dose for the pregnant participants (arm 1), and 0, 1 and 6 months for the non-pregnant participant (arm 3).
  Other Names: 26 kDa protein (239 amino acids, aa368 to aa606) encoded by ORF2 of the HEV1 (Chinese HEV strain, genotype 1) and is expressed in Escherichia coli as a non-fusion protein.
  Arms: Non-Pregnant participants receiving Hecolin®; Pregnant participant receiving Hecolin®
Other: Isotonic Sodium Chloride injection — Placebo will be administered 2 doses administered 4 weeks apart during pregnancy and 1 dose administered after delivery at least 20 weeks following the second dose for the pregnant participants (arm 2)
  Other Names: Sterile 0.9% sodium chloride
  Arms: Pregnant participants receiving placebo

SUMMARY:
This is a phase II randomized, observer-blinded, placebo-controlled study with 3 arms enrolling a total of 2,358 participants. The arms are composed of Arm 1, pregnant participants receiving Hecolin® (N=1,104) with immunogenicity subset (n=150), Arm 2, pregnant participants receiving placebo (N=1,104) with immunogenicity subset (n=150), and Arm 3, non-pregnant participants receiving Hecolin® (N=150) of which all participants in this arm will be included in the immunogenicity subset.

DETAILED DESCRIPTION:
Hecolin® is licensed in China and Pakistan indicated to be used for prevention of hepatitis E in healthy adult. The primary goal of this clinical trial is to establish the safety and immunogenicity of Hecolin® during pregnancy. As secondary and exploratory objectives, infant immune response through passive immunization of infants achieved through transplacental transfer of maternal IgG antibodies from the pregnant mother who has received Hecolin® in the second or third trimester will be evaluated.

Hecolin® follows a 3-dose schedule (0-1-6 months). For Arm 1 and 2, pregnant participants will receive 2 doses of Hecolin® or placebo at a 4 weeks interval and the third dose will be administered postpartum, approximately 20 weeks after the second dose. The neonates from these Arms will be followed for 24 weeks after birth. For Arm 3, non-pregnant participants will receive Hecolin® at 0-1-6 months schedule.

After each dose of IP injection to pregnant/non-pregnant participants, immediate AE (30 minutes post injection), solicited AE (7 days post injection), unsolicited AE (28 days post injection) and AESI/SAE (during the whole study period) will be collected.

For the immunogenicity subset, the participants' blood will be drawn before and 4 weeks post each dose of IP injection. At delivery, maternal blood will be drawn. Breast milk samples will be taken at delivery, 6 weeks, and 24 weekss after delivery.

All infant AESI/SAE will be collected throughout the study period and developmental assessment will be performed at age of 6 weeks, and 24 weeks. Blood will be drawn from infant immunogenicity subset at the same time points, umbilical cord blood (neonate blood will be collected if cord blood is not available for collection) at delivery, venous blood at age of 6 weeks and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a pregnant/non-pregnant woman must meet all of the following criteria:

Pregnant women only:

1. Healthy women 16-45 years of age who are between 14 0/7 and 34 6/7 weeks gestation1 on the day of planned vaccination with an uncomplicated, singleton pregnancy, who are at no known increased risk for complications for herself and her infant.
2. Individual willing to provide written informed consent for herself and her infant to participate in the study.
3. Individual who can be followed up during the study period and can comply with the study requirements.
4. Individual and fetus in good health as determined by the outcome of medical history, physical examination, obstetric history, prenatal care (by ultrasound and other prenatal assessment subject to gestational age), vital signs, laboratory evaluations at screening and the clinical judgment of the investigator.
5. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Non-pregnant women only:

1. Healthy women 16-45 years of age.
2. Individual willing to provide written informed consent to participate in the study.
3. Individual who can be followed up during the study period and can comply with the study requirements.
4. Individual in good health as determined by the outcome of medical history, physical examination, vital signs, laboratory evaluations at screening and the clinical judgment of the investigator.
5. Individuals who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
6. Females of childbearing potential with negative urinary pregnancy test on the day of screening.
7. Females of childbearing potential who are using an effective birth control method2 for at least 4 weeks before the screening and up to 4 weeks after the last vaccination.

Exclusion Criteria:

A pregnant/non-pregnant woman who meets any of the following criteria will be excluded from participation in this study:

1. Has received any hepatitis E vaccine in the past.
2. Febrile illness (axillary temperature ≥ 38.5°C) or acute illness within 3 days prior to the study vaccination.
3. Known history or allergy to study vaccine components and/or excipients or other medications, or any other allergies or medical history deemed by the investigator to increase the risk of an adverse event if they were to participate in the trial (e.g., Guillain-Barre Syndrome).
4. Major congenital abnormalities which in the opinion of investigator may affect the participant's participation in the study.
5. Known history of immune function disorders including immunodeficiency diseases (known HIV infection or other immune function disorders) and lupus.
6. Chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisone equivalent for periods exceeding 10 days), cytotoxic or other immunosuppressive drugs within past 6 weeks.
7. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the participant and interfere with the assessment of the study objectives.
8. Behavioral or cognitive impairment, or chronic substance abuse, or psychiatric disease or neural disorders, that, in the opinion of the investigator, could interfere with the participant's ability to participate in the trial.
9. History of splenectomy.
10. Past history of thrombocytopenia and/or thrombosis, myocarditis or pericarditis or any other significant cardiac condition.
11. With a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time resulting in contraindication for IM injections/blood extractions. (Those who receive low dose aspirin (less than 100mg/day) are not excluded)
12. Receipt of blood or blood-derived products in the past 3 months.
13. Receipt of other vaccines from 4 weeks prior to test vaccination or planned to receive any vaccine within 4 weeks of last dose of study vaccine
14. As per Investigator's medical judgement, an individual could be excluded from the study in spite of meeting all inclusion/exclusion criteria mentioned above.
15. Concomitantly enrolled or scheduled to be enrolled in another trial.
16. Research staff involved with the clinical study or family/household members of research staff.
17. Body mass index (BMI) of ≥ 40, at the time of the screening visit.

Pregnant women only:

1. Plans to terminate her pregnancy. Pregnancy complications (in the current pregnancy) such as preterm labor, gestational diabetes, hypertension (blood pressure (BP) > 140/90 in the presence of proteinuria or BP > 150/100 with or without proteinuria), or currently on an antihypertensive therapy, or pre-eclampsia, or evidence of intrauterine growth restriction.

3. Prior stillbirth or neonatal death, or multiple (≥ 3) spontaneous abortions. 4. Prior preterm delivery ≤ 34 weeks gestation or having ongoing intervention (medical/surgical) in current pregnancy to prevent preterm birth.

5. Previous infant with a known genetic disorder or major congenital anomaly. 6. History of major gynecologic or major abdominal surgery (previous Caesarean section is not an exclusion) 7. Current pregnancy results from in vitro fertilization (IVF). 8. Current pregnancy results from rape or incest. 9. Plans to release the neonate for adoption or the neonate to be a ward of the state.

10. Greater than 5 prior deliveries

Non-pregnant women only:

1. Pregnant or plan to be pregnant during the study period.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2358 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of pregnancy-related AESI and SAE from vaccination in pregnant participant. | Throughout the study period, approximately 24 months.
  * Proportion of pregnancy-related AESI from the vaccination throughout the entire study in pregnant participants.
  * Proportion of SAE from the vaccination throughout the entire study in pregnant participants.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post second dose of Hecolin®
  GMC of anti-HEV IgG at 4 weeks post second dose of Hecolin® administered 4 weeks apart in pregnant women and non-pregnant women.

SECONDARY OUTCOMES:
Proportion of AESIs and SAE in neonate/infant participants. | 6 months of life in neonate/infant
  * Proportion of neonatal/infant AESIs.
  * Proportion of SAE through the 6 months of life in neonate/infant.
Proportion of immediate adverse events in pregnant and non-pregnant participants | Within 30 minutes post each dose of vaccination.
  Proportion of immediate adverse events within 30 minutes post each dose of vaccination in pregnant and non-pregnant participants.
Proportion of Solicited local and system adverse events in pregnant and non-pregnant participants | Within 7 days post each dose of vaccination.
  Proportion of solicited local and systemic adverse events within 7 days post each dose of vaccination in pregnant and non-pregnant participants.
Proportion of unsolicited adverse events in pregnant and non-pregnant participants | Within 28 days post each dose of vaccination.
  Proportion of unsolicited adverse events within 28 days post each dose of vaccination in pregnant and non-pregnant participants.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post second dose of vaccination.
  SCR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post second dose of Hecolin® administered 4 weeks apart in pregnant and non-pregnant participants.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post third dose of vaccination.
  GMC of anti-HEV IgG at 4 weeks post third dose of Hecolin® (2 doses in pregnancy and 1 dose after delivery) in pregnant and non-pregnant participants.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post third dose of vaccination.
  SCR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post third dose of Hecolin® (2 doses in pregnancy and 1 dose after delivery) in pregnant and non-pregnant participants.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post first dose of vaccination.
  GMC of anti-HEV IgG at 4 weeks post first dose of Hecolin® in pregnant and non-pregnant participants.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post first dose of vaccination.
  SCR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post first dose of Hecolin® in pregnant and non-pregnant participants.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post second dose of vaccination.
  GMC of anti-HEV IgG at 4 weeks post second dose of Hecolin® in pregnant participants of GA 14-27 weeks (second trimester) and 28-34 weeks (third trimester) and non-pregnant participants as measured by anti HEV IgG ELISA.
Immunogenicity in pregnant and non-pregnant participants | 4 weeks post second dose of vaccination.
  SCR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post second dose of Hecolin® in pregnant participants of GA 14-27 weeks (second trimester) and 28-34 weeks (third trimester) and non-pregnant participants.

OTHER OUTCOMES:
Proportion of vaginal delivery, elective cesarian section and emergency cesarian section in pregnant participants. | throughout the study
Immunogenicity in neonate/infant participants | at delivery, infant age of 6 weeks and 6 months
  * GMC of anti-HEV IgG in neonates/infants at delivery and age of 6 weeks and 6 months.
  * Anti-HEV IgG Subclass
Immunogenicity in maternal blood and umbilical cord at delivery | at time of delivery
  * GMC of anti-HEV IgG in maternal blood and umbilical cord at the time of delivery
  * Anti-HEV IgG Subclass
Immunogenicity in breastmilk | at delivery, 6 weeks and 6 months post partum
  * GMC of anti-HEV IgG in breastmilk at delivery and postpartum 6 weeks and 6 months.
  * Anti-HEV IgG Subclass
Counts and proportion of laboratory confirmed Hepatitis E among pregnant recipients of Hecolin® and placebo and their infants during pregnancy and 6 months after birth. | throughout the study period, approximately 24 months
Safety in seropositive and seronegative pregnant participants at baseline | throughout the study period, approximately 24 months
  * Proportion of pregnancy-related AESI from the vaccination throughout the entire study in pregnant participants by serostatus.
  * Proportion of SAE from the vaccination throughout the entire study in pregnant by serostatus.
Immunogenicity in seropositive and seronegative pregnant and non-pregnant participants | 4 weeks post third dose of vaccination.
  GMC of anti-HEV IgG at 4 weeks post third dose of Hecolin® (2 doses in pregnancy and 1 dose after delivery) in pregnant and non-pregnant participants depending on serostatus.

CONTACTS AND LOCATIONS:
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonhoeffer J, Kochhar S, Hirschfeld S, Heath PT, Jones CE, Bauwens J, Honrado A, Heininger U, Munoz FM, Eckert L, Steinhoff M, Black S, Padula M, Sturkenboom M, Buttery J, Pless R, Zuber P; GAIA project participants. Global alignment of immunization safety assessment in pregnancy - The GAIA project. Vaccine. 2016 Dec 1;34(49):5993-5997. doi: 10.1016/j.vaccine.2016.07.006. Epub 2016 Oct 14. PMID 27751641
- [Result] Madhi SA, Polack FP, Piedra PA, Munoz FM, Trenholme AA, Simoes EAF, Swamy GK, Agrawal S, Ahmed K, August A, Baqui AH, Calvert A, Chen J, Cho I, Cotton MF, Cutland CL, Englund JA, Fix A, Gonik B, Hammitt L, Heath PT, de Jesus JN, Jones CE, Khalil A, Kimberlin DW, Libster R, Llapur CJ, Lucero M, Perez Marc G, Marshall HS, Masenya MS, Martinon-Torres F, Meece JK, Nolan TM, Osman A, Perrett KP, Plested JS, Richmond PC, Snape MD, Shakib JH, Shinde V, Stoney T, Thomas DN, Tita AT, Varner MW, Vatish M, Vrbicky K, Wen J, Zaman K, Zar HJ, Glenn GM, Fries LF; Prepare Study Group. Respiratory Syncytial Virus Vaccination during Pregnancy and Effects in Infants. N Engl J Med. 2020 Jul 30;383(5):426-439. doi: 10.1056/NEJMoa1908380. PMID 32726529
- [Result] Rein DB, Stevens GA, Theaker J, Wittenborn JS, Wiersma ST. The global burden of hepatitis E virus genotypes 1 and 2 in 2005. Hepatology. 2012 Apr;55(4):988-97. doi: 10.1002/hep.25505. PMID 22121109
- [Result] Beniwal M, Kumar A, Kar P, Jilani N, Sharma JB. Prevalence and severity of acute viral hepatitis and fulminant hepatitis during pregnancy: a prospective study from north India. Indian J Med Microbiol. 2003 Jul-Sep;21(3):184-5. PMID 17643015
- [Result] Kumar RM, Uduman S, Rana S, Kochiyil JK, Usmani A, Thomas L. Sero-prevalence and mother-to-infant transmission of hepatitis E virus among pregnant women in the United Arab Emirates. Eur J Obstet Gynecol Reprod Biol. 2001 Dec 10;100(1):9-15. doi: 10.1016/s0301-2115(01)00448-1. PMID 11728649
- [Result] Medhat A, el-Sharkawy MM, Shaaban MM, Makhlouf MM, Ghaneima SE. Acute viral hepatitis in pregnancy. Int J Gynaecol Obstet. 1993 Jan;40(1):25-31. doi: 10.1016/0020-7292(93)90768-r. PMID 8094346
- [Result] Patra S, Kumar A, Trivedi SS, Puri M, Sarin SK. Maternal and fetal outcomes in pregnant women with acute hepatitis E virus infection. Ann Intern Med. 2007 Jul 3;147(1):28-33. doi: 10.7326/0003-4819-147-1-200707030-00005. PMID 17606958
- [Result] Nelson KE, Heaney CD, Labrique AB, Kmush BL, Krain LJ. Hepatitis E: prevention and treatment. Curr Opin Infect Dis. 2016 Oct;29(5):478-85. doi: 10.1097/QCO.0000000000000294. PMID 27454402
- [Result] Aggarwal R. Clinical presentation of hepatitis E. Virus Res. 2011 Oct;161(1):15-22. doi: 10.1016/j.virusres.2011.03.017. Epub 2011 Mar 31. PMID 21458513
- [Result] Kamar N, Lhomme S, Abravanel F, Cointault O, Esposito L, Cardeau-Desangles I, Del Bello A, Dorr G, Lavayssiere L, Nogier MB, Guitard J, Ribes D, Goin AL, Broue P, Metsu D, Saune K, Rostaing L, Izopet J. An Early Viral Response Predicts the Virological Response to Ribavirin in Hepatitis E Virus Organ Transplant Patients. Transplantation. 2015 Oct;99(10):2124-31. doi: 10.1097/TP.0000000000000850. PMID 26214817
- [Result] Khuroo MS, Kamili S. Aetiology, clinical course and outcome of sporadic acute viral hepatitis in pregnancy. J Viral Hepat. 2003 Jan;10(1):61-9. doi: 10.1046/j.1365-2893.2003.00398.x. PMID 12558914
- [Result] Holla RP, Ahmad I, Ahmad Z, Jameel S. Molecular virology of hepatitis E virus. Semin Liver Dis. 2013 Feb;33(1):3-14. doi: 10.1055/s-0033-1338110. Epub 2013 Apr 5. PMID 23564385
- [Result] Mori Y, Matsuura Y. Structure of hepatitis E viral particle. Virus Res. 2011 Oct;161(1):59-64. doi: 10.1016/j.virusres.2011.03.015. Epub 2011 Apr 1. PMID 21440590
- [Result] Iqbal M, Ahmed A, Qamar A, Dixon K, Duncan JF, Islam NU, Rauf A, Bryan JP, Malik IA, Legters LJ. An outbreak of enterically transmitted non-A, non-B hepatitis in Pakistan. Am J Trop Med Hyg. 1989 Apr;40(4):438-43. doi: 10.4269/ajtmh.1989.40.438. PMID 2496611
- [Result] Butt AS, Sharif F. Viral Hepatitis in Pakistan: Past, Present, and Future. Euroasian J Hepatogastroenterol. 2016 Jan-Jun;6(1):70-81. doi: 10.5005/jp-journals-10018-1172. Epub 2016 Jul 9. PMID 29201731
- [Result] Jin H, Zhao Y, Zhang X, Wang B, Liu P. Case-fatality risk of pregnant women with acute viral hepatitis type E: a systematic review and meta-analysis. Epidemiol Infect. 2016 Jul;144(10):2098-106. doi: 10.1017/S0950268816000418. Epub 2016 Mar 4. PMID 26939626
- [Result] Hakim MS, Wang W, Bramer WM, Geng J, Huang F, de Man RA, Peppelenbosch MP, Pan Q. The global burden of hepatitis E outbreaks: a systematic review. Liver Int. 2017 Jan;37(1):19-31. doi: 10.1111/liv.13237. Epub 2016 Sep 9. PMID 27542764
- [Result] Scott RM, Kmush BL, Norkye K, Hada M, Shrestha MP, Vaughn DW, Myint KSA, Endy TP, Shrestha SK, Innis BL. Historical Analysis of the Risk of Hepatitis E and Its Complications in Pregnant Women in Nepal, 1996-1998. Am J Trop Med Hyg. 2021 Jun 14;105(2):440-448. doi: 10.4269/ajtmh.20-1007. PMID 34125701
- [Result] Gurley ES, Halder AK, Streatfield PK, Sazzad HM, Huda TM, Hossain MJ, Luby SP. Estimating the burden of maternal and neonatal deaths associated with jaundice in Bangladesh: possible role of hepatitis E infection. Am J Public Health. 2012 Dec;102(12):2248-54. doi: 10.2105/AJPH.2012.300749. Epub 2012 Oct 18. PMID 23078501
- [Result] Labrique AB, Sikder SS, Krain LJ, West KP Jr, Christian P, Rashid M, Nelson KE. Hepatitis E, a vaccine-preventable cause of maternal deaths. Emerg Infect Dis. 2012 Sep;18(9):1401-4. doi: 10.3201/eid1809.120241. PMID 22931753
- [Result] Khuroo MS. Hepatitis E and Pregnancy: An Unholy Alliance Unmasked from Kashmir, India. Viruses. 2021 Jul 9;13(7):1329. doi: 10.3390/v13071329. PMID 34372535
- [Result] Bigna JJ, Modiyinji AF, Nansseu JR, Amougou MA, Nola M, Kenmoe S, Temfack E, Njouom R. Burden of hepatitis E virus infection in pregnancy and maternofoetal outcomes: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2020 Jul 28;20(1):426. doi: 10.1186/s12884-020-03116-2. PMID 32723309
- [Result] Puri M, Patra S, Singh P, Malhotra N, Trivedi SS, Sharma S, Kumar A, Sarin SK. Factors influencing occurrence of postpartum haemorrhage in pregnant women with hepatitis E infection and deranged coagulation profile. Obstet Med. 2011 Sep;4(3):108-12. doi: 10.1258/om.2011.110031. Epub 2011 Aug 23. PMID 27579103
- [Result] Krain LJ, Atwell JE, Nelson KE, Labrique AB. Fetal and neonatal health consequences of vertically transmitted hepatitis E virus infection. Am J Trop Med Hyg. 2014 Feb;90(2):365-70. doi: 10.4269/ajtmh.13-0265. Epub 2014 Jan 13. PMID 24420778
- [Result] Khuroo MS, Kamili S, Khuroo MS. Clinical course and duration of viremia in vertically transmitted hepatitis E virus (HEV) infection in babies born to HEV-infected mothers. J Viral Hepat. 2009 Jul;16(7):519-23. doi: 10.1111/j.1365-2893.2009.01101.x. Epub 2009 Feb 17. PMID 19228284
- [Result] Sharma S, Kumar A, Kar P, Agarwal S, Ramji S, Husain SA, Prasad S, Sharma S. Risk factors for vertical transmission of hepatitis E virus infection. J Viral Hepat. 2017 Nov;24(11):1067-1075. doi: 10.1111/jvh.12730. Epub 2017 Jul 12. PMID 28570034
- [Result] Berglov A, Hallager S, Weis N. Hepatitis E during pregnancy: Maternal and foetal case-fatality rates and adverse outcomes-A systematic review. J Viral Hepat. 2019 Nov;26(11):1240-1248. doi: 10.1111/jvh.13129. Epub 2019 Jun 14. PMID 31095813
- [Result] Jilani N, Das BC, Husain SA, Baweja UK, Chattopadhya D, Gupta RK, Sardana S, Kar P. Hepatitis E virus infection and fulminant hepatic failure during pregnancy. J Gastroenterol Hepatol. 2007 May;22(5):676-82. doi: 10.1111/j.1440-1746.2007.04913.x. PMID 17444855
- [Result] Ratho RK, Thakur V, Arya S, Singh MP, Suri V, Das A. Placenta as a site of HEV replication and inflammatory cytokines modulating the immunopathogenesis of HEV in pregnant women. J Med Virol. 2022 Jul;94(7):3457-3463. doi: 10.1002/jmv.27699. Epub 2022 Mar 24. PMID 35257382
- [Result] Gouilly J, Chen Q, Siewiera J, Cartron G, Levy C, Dubois M, Al-Daccak R, Izopet J, Jabrane-Ferrat N, El Costa H. Genotype specific pathogenicity of hepatitis E virus at the human maternal-fetal interface. Nat Commun. 2018 Nov 12;9(1):4748. doi: 10.1038/s41467-018-07200-2. PMID 30420629
- [Result] Zaman K, Dudman S, Stene-Johansen K, Qadri F, Yunus M, Sandbu S, Gurley ES, Overbo J, Julin CH, Dembinski JL, Nahar Q, Rahman A, Bhuiyan TR, Rahman M, Haque W, Khan J, Aziz A, Khanam M, Streatfield PK, Clemens JD. HEV study protocol : design of a cluster-randomised, blinded trial to assess the safety, immunogenicity and effectiveness of the hepatitis E vaccine HEV 239 (Hecolin) in women of childbearing age in rural Bangladesh. BMJ Open. 2020 Jan 19;10(1):e033702. doi: 10.1136/bmjopen-2019-033702. PMID 31959609
- [Result] Wu T, Zhu FC, Huang SJ, Zhang XF, Wang ZZ, Zhang J, Xia NS. Safety of the hepatitis E vaccine for pregnant women: a preliminary analysis. Hepatology. 2012 Jun;55(6):2038. doi: 10.1002/hep.25522. No abstract available. PMID 22161542
- [Result] Zhu FC, Zhang J, Zhang XF, Zhou C, Wang ZZ, Huang SJ, Wang H, Yang CL, Jiang HM, Cai JP, Wang YJ, Ai X, Hu YM, Tang Q, Yao X, Yan Q, Xian YL, Wu T, Li YM, Miao J, Ng MH, Shih JW, Xia NS. Efficacy and safety of a recombinant hepatitis E vaccine in healthy adults: a large-scale, randomised, double-blind placebo-controlled, phase 3 trial. Lancet. 2010 Sep 11;376(9744):895-902. doi: 10.1016/S0140-6736(10)61030-6. Epub 2010 Aug 20. PMID 20728932
- [Result] Qiao YL, Wu T, Li RC, Hu YM, Wei LH, Li CG, Chen W, Huang SJ, Zhao FH, Li MQ, Pan QJ, Zhang X, Li Q, Hong Y, Zhao C, Zhang WH, Li YP, Chu K, Li M, Jiang YF, Li J, Zhao H, Lin ZJ, Cui XL, Liu WY, Li CH, Guo DP, Ke LD, Wu X, Tang J, Gao GQ, Li BY, Zhao B, Zheng FX, Dai CH, Guo M, Zhao J, Su YY, Wang JZ, Zhu FC, Li SW, Pan HR, Li YM, Zhang J, Xia NS. Efficacy, Safety, and Immunogenicity of an Escherichia coli-Produced Bivalent Human Papillomavirus Vaccine: An Interim Analysis of a Randomized Clinical Trial. J Natl Cancer Inst. 2020 Feb 1;112(2):145-153. doi: 10.1093/jnci/djz074. PMID 31086947
- [Result] Aye TT, Uchida T, Ma XZ, Iida F, Shikata T, Zhuang H, Win KM. Complete nucleotide sequence of a hepatitis E virus isolated from the Xinjiang epidemic (1986-1988) of China. Nucleic Acids Res. 1992 Jul 11;20(13):3512. doi: 10.1093/nar/20.13.3512. No abstract available. PMID 1630924
- [Result] Li SW, Zhang J, He ZQ, Gu Y, Liu RS, Lin J, Chen YX, Ng MH, Xia NS. Mutational analysis of essential interactions involved in the assembly of hepatitis E virus capsid. J Biol Chem. 2005 Feb 4;280(5):3400-6. doi: 10.1074/jbc.M410361200. Epub 2004 Nov 22. PMID 15557331
- [Result] Wei M, Zhang X, Yu H, Tang ZM, Wang K, Li Z, Zheng Z, Li S, Zhang J, Xia N, Zhao Q. Bacteria expressed hepatitis E virus capsid proteins maintain virion-like epitopes. Vaccine. 2014 May 19;32(24):2859-65. doi: 10.1016/j.vaccine.2014.02.025. Epub 2014 Mar 22. PMID 24662711
- [Result] Li SW, Zhang J, Li YM, Ou SH, Huang GY, He ZQ, Ge SX, Xian YL, Pang SQ, Ng MH, Xia NS. A bacterially expressed particulate hepatitis E vaccine: antigenicity, immunogenicity and protectivity on primates. Vaccine. 2005 Apr 22;23(22):2893-901. doi: 10.1016/j.vaccine.2004.11.064. PMID 15780738
- [Result] Zhang J, Liu CB, Li RC, Li YM, Zheng YJ, Li YP, Luo D, Pan BB, Nong Y, Ge SX, Xiong JH, Shih JW, Ng MH, Xia NS. Randomized-controlled phase II clinical trial of a bacterially expressed recombinant hepatitis E vaccine. Vaccine. 2009 Mar 13;27(12):1869-74. doi: 10.1016/j.vaccine.2008.12.061. Epub 2009 Jan 23. PMID 19168109
- [Result] Zhang J, Zhang XF, Huang SJ, Wu T, Hu YM, Wang ZZ, Wang H, Jiang HM, Wang YJ, Yan Q, Guo M, Liu XH, Li JX, Yang CL, Tang Q, Jiang RJ, Pan HR, Li YM, Shih JW, Ng MH, Zhu FC, Xia NS. Long-term efficacy of a hepatitis E vaccine. N Engl J Med. 2015 Mar 5;372(10):914-22. doi: 10.1056/NEJMoa1406011. PMID 25738667
- [Result] Tavares Da Silva F, Gonik B, McMillan M, Keech C, Dellicour S, Bhange S, Tila M, Harper DM, Woods C, Kawai AT, Kochhar S, Munoz FM; Brighton Collaboration Stillbirth Working Group. Stillbirth: Case definition and guidelines for data collection, analysis, and presentation of maternal immunization safety data. Vaccine. 2016 Dec 1;34(49):6057-6068. doi: 10.1016/j.vaccine.2016.03.044. Epub 2016 Jul 16. No abstract available. PMID 27431422
- [Result] Pathirana J, Munoz FM, Abbing-Karahagopian V, Bhat N, Harris T, Kapoor A, Keene DL, Mangili A, Padula MA, Pande SL, Pool V, Pourmalek F, Varricchio F, Kochhar S, Cutland CL; Brighton Collaboration Neonatal Death Working Group. Neonatal death: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016 Dec 1;34(49):6027-6037. doi: 10.1016/j.vaccine.2016.03.040. Epub 2016 Jul 19. PMID 27449077
- [Result] Jones CE, Munoz FM, Kochhar S, Vergnano S, Cutland CL, Steinhoff M, Black S, Heininger U, Bonhoeffer J, Heath PT. Guidance for the collection of case report form variables to assess safety in clinical trials of vaccines in pregnancy. Vaccine. 2016 Dec 1;34(49):6007-6014. doi: 10.1016/j.vaccine.2016.07.007. Epub 2016 Oct 25. PMID 27793485
- [Result] Bendall R, Ellis V, Ijaz S, Ali R, Dalton H. A comparison of two commercially available anti-HEV IgG kits and a re-evaluation of anti-HEV IgG seroprevalence data in developed countries. J Med Virol. 2010 May;82(5):799-805. doi: 10.1002/jmv.21656. PMID 20336757
- [Result] Stout MJ, Busam R, Macones GA, Tuuli MG. Spontaneous and indicated preterm birth subtypes: interobserver agreement and accuracy of classification. Am J Obstet Gynecol. 2014 Nov;211(5):530.e1-4. doi: 10.1016/j.ajog.2014.05.023. Epub 2014 May 17. PMID 24844852
- [Result] Fulton TR, Narayanan D, Bonhoeffer J, Ortiz JR, Lambach P, Omer SB. A systematic review of adverse events following immunization during pregnancy and the newborn period. Vaccine. 2015 Nov 25;33(47):6453-65. doi: 10.1016/j.vaccine.2015.08.043. Epub 2015 Sep 26. PMID 26413879